CLINICAL TRIAL: NCT01723527
Title: Diversion to Treatment for Injection Drug Users Arrested for Possession of Heroin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Anthony DeFulio, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA033510-01 (NIH)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Cocaine-Related Disorders; HIV; Heroin Dependence
Keywords: Cocaine; Heroin; HIV; Contingency Management; Incentives; Criminal Justice; Methadone; Buprenorphine; Employment; Job Training; Wage Subsidies
MeSH Terms: conditions — Cocaine-Related Disorders; Heroin Dependence | interventions — Methadone; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Workplace (Experimental): Participants assigned to this condition will receive the standard services and requirements for diversion as described for the usual care group, and will also be eligible to attend the three-phase Therapeutic Workplace (TW) intervention. All phases of this intervention include employment-based drug abstinence reinforcement contingencies. Under these contingencies, participants can work and earn wages or wage subsidies contingent upon drug abstinence as verified by urinalysis. Phase 1 of the TW intervention is expected to increase cocaine abstinence and to prepare participants for employment. Phase 2 of the TW intervention is expected to maintain abstinence while participants are employed in an onsite model workplace. Phase 3 is designed to increase employment in community jobs and to maintain abstinence while participants are employed in offsite community workplaces.
  Interventions: Drug: Methadone; Drug: Buprenorphine; Behavioral: Employment-based drug abstinence reinforcement
- Diversion to treatment (Usual Care) (Active Comparator): Participants in this condition will be offered the standard treatment services available in community methadone and buprenorphine programs, including medication (methadone or buprenorphine, respectively), counseling services, HIV testing, and case management. All services will be provided in the treatment clinics. There are a number of clinics within easy walking distance from the research site, and others throughout the city that are reachable by public transportation from the research site. In addition, all participants will receive referrals to the Re-Entry Center, a One-Stop Career Center tailored to the needs of offenders, at all intake and monthly assessments. As mentioned in detail above, participants will be required by the court to stay enrolled in treatment for 90 days. It is important to note that all diverted individuals will receive these services and requirements, independent of whether they agree to participate in the pilot study.
  Interventions: Drug: Methadone; Drug: Buprenorphine

INTERVENTIONS:
Drug: Methadone — Clinic-Based Methadone Maintenance Treatment
Drug: Buprenorphine — Clinic-Based Buprenorphine Maintenance Treatment
Behavioral: Employment-based drug abstinence reinforcement
  Other Names: Therapeutic Workplace
  Arms: Therapeutic Workplace

SUMMARY:
More Americans are arrested for drug offenses than for any other crime. In 2009, over 294,000 arrests were made for possession of cocaine or heroin. Incarceration does not address the root problems and is frequently followed by relapse and re-arrest after release. In the case of opiate-dependent adults arrested for possession of heroin, one potentially effective alternative is to divert offenders to methadone maintenance treatment (MMT) as an alternative to adjudication of their case. MMT is an effective treatment for heroin dependence, and appears very effective for criminal offenders. However, cocaine use is common in MMT patients, including those with recent criminal justice involvement, and MMT alone is ineffective in addressing cocaine use. Continued cocaine use carries a substantial health burden and necessarily entails continued criminal activity. Thus, treatment for diverted opiate-dependent offenders should be designed to address cocaine use as well as opiate use. A Stage 1 Behavior Therapy Development project is planned over 2 years to adapt, manualize and pilot test the Therapeutic Workplace intervention for adults charged with heroin possession and offered diversion to methadone maintenance treatment as an alternative to adjudication of their case. The Therapeutic Workplace is a novel, employment-based contingency management intervention that has been very effective in promoting cocaine abstinence in adults who use cocaine persistently during methadone treatment. In the Therapeutic Workplace, participants are hired in a model workplace and required to provide drug-free urine samples to work and to earn maximum pay. Once we develop and manualize the adapted version of the Therapeutic Workplace for adults arrested for heroin possession, a pilot test will be conducted. Individuals identified by the State Attorney's office as candidates for diversion will be assessed for study eligibility. Given the high rates of injection drug use and injection-related transmission of HIV in Baltimore, this study will be restricted to injection drug users to evaluate the potential utility of this intervention in reducing HIV risk. Eligible individuals will be offered methadone maintenance in lieu of prosecution and will be required to remain in methadone treatment for 90 days. All participants will receive standard MMT, independent of whether they decide to participate in the pilot study. After beginning MMT, participants will be invited to enroll in the pilot study and randomly assigned to two study groups. Participants assigned to the Usual Care Diversion group will receive the standard MMT. Participants assigned to the Therapeutic Workplace Enhanced Diversion group will receive the standard MMT and the Therapeutic Workplace intervention. The data from this pilot study will serve as the foundation for a full-scaled randomized controlled trial. Overall, the Therapeutic Workplace could serve as a novel and ideal intervention for many heroin dependent adults involved in the criminal justice system. The use of MMT in lieu of adjudication in combination with the Therapeutic Workplace could increase drug abstinence and employment and decrease HIV risk and criminal activity in this refractory high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* report using heroin at least 20 of the last 30 days of living in the community
* meet criteria for methadone maintenance (at least one year of meeting DSM IV criteria for heroin dependence)
* have visible track marks or other clear physical evidence of injection drug use
* report using cocaine in the last 30 days
* were unemployed prior to arrest
* have a income below the federal poverty level
* live in the Baltimore City area

Exclusion Criteria:

* report current suicidal ideation or hallucinations
* receiving opioid pharmacotherapy prior to arrest
* have a serious uncontrolled medical condition that would prevent attendance in methadone or buprenorphine treatment
* are pregnant or breastfeeding
* have a physical imparement that would prevent typing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Cocaine abstinence as assessed by urinalysis | One year
  dichotomous (Y/N)
Cocaine abstinence as assessed by self-reports | One year
  dichotomous (Y/N)

SECONDARY OUTCOMES:
Any drug use (Y/N) | One year
  Any drug use will be counted as Yes if a urine sample indicates that the participant is positive for any of the DOT 5 drugs, or if the participant reports using any of the DOT 5 drugs (Amphetamines, Cocaine, Marijuana, Opiates, PCP).
Any engagement in HIV risk behavior (Y/N) | One year
  Any engagement in HIV risk behavior will be counted as Yes if a participant reports any unprotected vaginal or anal sex or reports any injection drug use that includes the sharing of injection equipment.
Any criminal activity (Y/N) | One year
  Criminal activity will counted as Yes if a participant reports any days of illegal activity in the previous 30 days, or has been arrested for any new crime in the previous 30 days according to publically available records maintained by the Maryland DPSCS.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DeFulio, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Learning and Health, Baltimore, Maryland, United States